CLINICAL TRIAL: NCT05860010
Title: Comparing the Hemodynamic Effects of Epinephrine Versus Dexmedetomidine as an Adjuvant to Bupivacaine in Caudal Anaesthesia Assessed by Cardiometry: a Randomized, Double-blind, Controlled Study
Brief Title: Comparing the Hemodynamic Effects of Epinephrine Versus Dexmedetomidine as an Adjuvant to Bupivacaine in Caudal Anaesthesia Assessed by Cardiometry
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ayman Abougabal, consultant of anesthesia, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MD-375-2020
Record Dates: First submitted 2023-03-04; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Anesthesia, Local
MeSH Terms: interventions — Epinephrine; Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (Placebo Comparator): Bupivacaine will be administered in the caudal space
  Interventions: Drug: Bupivacaine
- dexmedetomidine (Active Comparator): caudal with dexmedetomidine
  Interventions: Drug: Dexmedetomidine; Drug: Bupivacaine
- epinephrine (Active Comparator): caudal with epinephrine
  Interventions: Drug: Epinephrine injection; Drug: Bupivacaine

INTERVENTIONS:
Drug: Epinephrine injection — patients will be placed on left lateral position and drug will be given the caudal space
  Arms: epinephrine
Drug: Dexmedetomidine — patients will be placed on left lateral position and drug will be given the caudal space
  Arms: dexmedetomidine
Drug: Bupivacaine — patients will be placed on left lateral position and drug will be given the caudal space

SUMMARY:
Electrical cardiometry (EC) is a non-invasive method of estimating cardiac parameters by measuring changes in thoracic bioimpedance during the cardiac cycle. The ICON (Cardiotronic Osypka Medical, San Diego, California) monitor uses four electrocardiogram electrodes and estimates the maximum rate of impedance change to peak aortic blood acceleration. An impedance change occurs between diastole and systole as red blood cell orientation is altered from random during diastole to align during systole. This device is validated against Fick cardiac output and transthoracic echocardiography in infants and children, as well as thermodilution in adults with R values of 0.9. This device is approved by the Food and Drug Administration (FDA) for use in pediatrics. Hypotension is expected to occur after epidural anesthesia (EA) due to the dilatation of venous vessels by sympathetic blockade with a subsequent decrease in venous return and cardiac output (CO). Also, the association of general anesthesia (GA) to EA can lead to more decrease in CO. The addition of epinephrine to local anesthetics (LA) could worsen hypotension through the systemic absorption of epinephrine that leads to a vasodilator β effect. Yet, CO may be enhanced by this β-adrenergic stimulation. However, it is well known that caudal epidural anesthesia has few or no hemodynamic changes in children less than 8 yr old. This could be attributed to the immaturity of their sympathetic system and smaller lower-limbs blood volume compared to adults. Caudal anesthesia is highly effective in abdominal, urinary tract, and lower extremity surgeries in children for intra- and postoperative analgesia. The addition of dexmedetomidine to local anesthetics in caudal anesthesia is a frequent practice. Dexmedetomidine, a highly selective alpha-2 adrenoreceptor agonist, is used as an intravenous sedative and analgesic drug. It has an a2/a1 selectivity ratio of 1600: 1 and is eight times more potent than clonidine. Intrathecal and epidural dexmedetomidine have been reported to produce analgesic properties, prolonging the duration of local anesthetics without causing nerve damage in pediatric patients.

Although basal heart rate is greater than in adults, activation of the parasympathetic nervous system, anesthetic overdose, or hypoxia can quickly trigger bradycardia and profound reductions in cardiac output. The sympathetic nervous system and baroreceptor reflexes are not fully mature and the infant cardiovascular system displays a blunted response to exogenous catecholamines. That's why it is very essential to determine the hemodynamic effects of any drug used as an adjuvant to local anesthetics for caudal block and to explore whether it reduces the child cardiac output or not.

As invasive cardiac monitors are rarely indicated in pediatric patients, and little is known about the impact of caudally administered dexmedetomidine on cardiac function, so we aimed to investigate its effect on hemodynamic functions measured by EC.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I and II, pediatric patients aged between 6 months and 8 years, of male or female gender, and undergoing elective infraumbilical (i.e. lower abdominal or genitourinary surgeries) will be included.

Exclusion Criteria:

* Parent or guardian refusal
* Patients < 6 months and > 8 years old
* Emergency cases
* Surgery lasting > 60 min
* Patients with known congenital heart disease.
* Patients with history or evidence of infection at the back.
* Congenital abnormalities of lower spine or meninges e.g. spina bifida
* Patients with blood clotting disorders or on anticoagulation therapy.
* Patients with known allergy to systemic or local anesthetics

Ages: 2 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Estimated)
Dates: Start 2023-06-05 (Estimated); Primary Completion 2023-11-05 (Estimated); Study Completion 2023-12-05 (Estimated)

PRIMARY OUTCOMES:
The percentage change in cardiac output after caudal injection | 15 minutes after caudal injection
  the change of cardiac output before and after caudal injection in percent

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Ayman Abougabal [aabougabal], Cairo
  - Kasr Al Ainy, Cairo

IPD SHARING:
Plan to Share IPD: Yes